CLINICAL TRIAL: NCT04366271
Title: Phase II Clinical Trial to Explore the Efficacy of Allogeneic Mesenchymal Cells From Umbilical Cord Tissue in Patients With Severe Pulmonary Involvement by COVID-19
Brief Title: Clinical Trial of Allogeneic Mesenchymal Cells From Umbilical Cord Tissue in Patients With COVID-19
Acronym: MESCEL-COVID19
Status: Withdrawn | Phase: Phase 2 | Type: Interventional
Why Stopped: Lack of funding
Sponsor: Hospital Infantil Universitario Niño Jesús, Madrid, Spain (Other)
Collaborators: Apices Soluciones S.L. (Industry)
Responsible Party: Principal Investigator, Mrs. Laura Aranzasti, Dr, Hospital Infantil Universitario Niño Jesús, Madrid, Spain
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: MESCEL-COVID19; 2020-001450-22 (EudraCT Number)
Record Dates: First submitted 2020-04-23; First posted 2020-04-28 (Actual); Last update posted 2021-08-27 (Actual); Status verified 2021-08

CONDITIONS: COVID
Keywords: COVID-19; mesenchymal cells from umbilical cord
MeSH Terms: conditions — COVID-19 | interventions — Standard of Care

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Mesenchymal cells (Experimental): Undifferentiated allogeneic mesenchymal cells derived from umbilical cord tissue
  Interventions: Biological: Mesenchymal cells
- Standard of care (Active Comparator): Standard of care
  Interventions: Drug: Standard of care

INTERVENTIONS:
Biological: Mesenchymal cells — 1 infusion of undifferentiated allogeneic mesenchymal cells derived from umbilical cord tissue
  Arms: Mesenchymal cells
Drug: Standard of care — Best treatment option for COVID-19 according to investigator criteria
  Arms: Standard of care

SUMMARY:
The disease caused by the SARS-CoV-2 virus is a viral disease that infects the lungs, producing flu-like symptoms. Elderly infected patients and/or those with co-morbidities may suffer from acute respiratory distress syndrome due to pneumonia (COVID-19 disease). Given the high transmission, this virus has spread in recent months from Wuhan (China) to the whole world, becoming a global emergency pandemic. The lack of curative treatment for this disease justifies the need to carry out clinical trials that provide quality evidence on treatment options. Given the pathophysiology of the disease, which involves an uncontrolled inflammatory response of alveolar cells, a treatment that attenuates the cytokine cascade could be key in rescuing the patient's lung tissue. Mesenchymal cells, due to their immunoregulatory potential and regenerative capacity, can be an effective treatment for patients infected with the SARS-CoV-2 virus.

In the present study we propose a therapy with undifferentiated allogeneic mesenchymal cells derived from umbilical cord tissue, a treatment whose safety has already been described in other clinical trials and that shows promising results in pilot studies carried out in China.

ELIGIBILITY:
Inclusion Criteria:

1. Patients aged between 40 and 80 years
2. Body weight between 50 kg and 100 kg
3. PCR diagnosis of SARS-CoV-2 virus infection
4. Clinical diagnosis of severe lung involvement associated with SARSCoV- 2 virus infection according to the criteria of the National Health Commission of China, that is, patients who meet at least one of the following criteria:

   1. Respiratory distress with ≥ 30 breaths per minute; or
   2. Oxygen saturation ≤ 93% at baseline; or
   3. Partial arterial oxygen pressure (PaO2) / Fraction of inspiration of O2 (FiO2) ≤300mmHg. (PaO2 / FiO2 is accepted based on SatO2). Patients who do not require respiratory support, or who require noninvasive respiratory support (conventional, high-flow oxygen therapy, or non-invasive mechanical ventilation) are considered eligible.
5. Patients who are already receiving the standard medical treatment available for severe lung involvement associated with SARS-CoV-2 virus infection or any of the standard treatments are contraindicated in the patient and cannot be used and it is necessary to consider other alternatives.
6. Women who are surgically sterile or postmenopausal or women of childbearing potential with negative urine or serum pregnancy test or men willing to use condoms for the entire duration of the study or for three months after the last dose of the investigational drug, whichever is later, or have a partner who is using a contraceptive method with high efficacy, such as described above.
7. Signed informed consent.

Exclusion Criteria:

1. Clinical diagnosis of critically serious lung involvement associated with SARS-CoV-2 virus infection according to the criteria of the National Health Commission of China, that is, patients who meet any of the following criteria:

   1. Respiratory failure requiring invasive mechanical ventilation; or
   2. Shock; or
   3. Combination with failure of another organ; need for ICU admission for monitoring / treatment.
2. Patients who are expected to develop rapidly fatal disease within 72 hours of enrollment.
3. Inability to maintain a mean arterial pressure > 50 mmHg before selection despite the presence of vasopressors and intravenous fluids.
4. Patients requiring treatment with vasopressors (dopamine > 5 mg / kg / min or any dose of epinephrine, norepinephrine, phenylephrine, or vasopressin) for at least 2 hours to maintain systolic blood pressure (SBP) > 90 mmHg (or mean blood pressure [MBP] > 70 mmHg) after adequate fluid administration.
5. Patients who are not expected to live more than 3 months due to other medical illnesses, such as neoplasia or other terminal illnesses.
6. Patients with primary or metastatic lung cancer or with chemotherapy scheduled for the next 90 days.
7. Patients with a known primary immunodeficiency disorder or with acquired immunodeficiency syndrome (HIV infection) with a CD4 count <200 cells / mm3 or who do not have an undetectable viral load (<200 copies).
8. Patients receiving immunosuppressive therapy (including chronic treatment with any alpha antitumor necrosis factor [TNFa]) or corticosteroid therapy.
9. Granulocytopenia, not due to sepsis, evidenced by an absolute neutrophil count <500 per μL.
10. Hematologic or lympho-reticular malignancies, unless in remission.
11. Patients who have received a stem cell, organ, or bone marrow transplant in the last 6 months.
12. Patients in current treatment with a biological product (eg, antibodies, cell therapy) or with plasmapheresis in the last 8 weeks.
13. Patients who are currently receiving or have received another investigational drug in the 90 days prior to study initiation (or 5 halflives of the investigational compound, whichever is longer).
14. Known allergies or hypersensitivity to antibiotics and/or any component of the investigational product.
15. Patients with known severe liver function impairment.
16. Patients with known severe kidney function impairment.
17. Patients admitted in the previous 15 days for causes other than SARS-CoV-2 virus infection.
18. Diseases other than SARS-CoV-2 virus infection leading to New York Heart Association class IV status.
19. Terminal neuromuscular disorders that alter the gradual withdrawal of the ventilator (eg, amyotrophic lateral sclerosis).
20. Patients with complete tetraplegia (traumatic or otherwise).
21. Dementia-Alzheimer and another situation in which is considered patient can not understand what is explaining, can not read or does not understand the language.

Ages: 40 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2020-05-07 (Actual); Primary Completion 2020-07-31 (Actual); Study Completion 2021-05-31 (Actual)

PRIMARY OUTCOMES:
Mortality due to lung involvement due to SARS-CoV-2 virus infection at 28 days of treatment | 28 days
  Percentage of patients death due to lung involvement due to SARS-CoV-2 virus infection at 28 days of treatment

SECONDARY OUTCOMES:
Mortality due to lung involvement due to SARS-CoV-2 virus infection at 14 days of treatment | 14 days
  Percentage of patients death due to lung involvement due to SARS-CoV-2 virus infection at 14 days of treatment
Mortality from any cause at 28 days | 28 days
  Percentage of patients death due to any cause at 28 days of treatment
Days without mechanical respirator and without vasopressor treatment for 28 days | 28 days
  Number of days without mechanical respirator and without vasopressor treatment for 28 days
Patients alive without mechanical ventilation and without vasopressors on day 28 | 28 days
  Percentage of patients alive without mechanical ventilation and without vasopressors on day 28
Patients alive and without mechanical ventilation on day 14 | 14 days
  Percentage of patients alive and without mechanical ventilation on day 14
Patients alive and without mechanical ventilation on day 28 | 28 days
  Percentage of patients alive and without mechanical ventilation on day 28
Patients alive and without vasopressors on day 28 | 28 days
  Percentage of patients alive and without vasopressors on day 28
Days without vasopressors for 28 days | 28 days
  Number of days without vasopressors for 28 days
Patients cured at 15 days | 15 days
  Percentage of patients cured at 15 days
Incidence of Treatment-Emergent Adverse Events | 1 year
  Percentage of patients with each adverse event

CONTACTS AND LOCATIONS:
Overall Officials: Luis Madero, MD, Study Chair — Hospital Infantil Universitario Niño Jesús, Oncohematology Department
Locations (6):
- Spain (6):
  - Hospital Universitario de Getafe, Getafe, Madrid
  - Hospital Universitario de Cruces, Barakaldo
  - Hospital Universitario de La Princesa, Madrid
  - Hospital Infantil Universitario Niño Jesus, Madrid
  - Hospital Ramón Y Cajal, Madrid
  - Complejo Universitario La Paz, Madrid

IPD SHARING:
Plan to Share IPD: Undecided